CLINICAL TRIAL: NCT06311513
Title: Multi-Center Pilot Study to Evaluate Concentrated Bone Marrow Aspirate (cBMA) as a Treatment to Modify Post-Traumatic Osteoarthritis (PTOA) Following Revision Anterior Cruciate Ligament Reconstruction (ACLR)
Brief Title: Concentrated Bone Marrow Aspirate in Revision ACL Reconstruction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Emory University (Other); Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-1017; 1177535 (Other Grant/Funding Number: Arthritis Foundation)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Anterior Cruciate Ligament Injuries; Post-Traumatic Osteoarthritis of Knee; Bone Marrow Aspirate Concentrate; ACL Injury
Keywords: Regenerative Medicine; Orthobiologics; Concentrated Bone Marrow Aspirate; Revision ACLR
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: This is a single-blinded randomized controlled trial. Participants will be allocated to either:
  1. Investigational arm (Revision ACLR + cBMA)
  2. Control arm (Revision ACLR + Sham Incision)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Investigational Arm (Experimental): Patients undergoing revision anterior cruciate ligament reconstruction surgery will get an intraoperative injection of concentrated bone marrow aspirate (cBMA).
  Interventions: Biological: Concentrated Bone Marrow Aspirate Injection; Procedure: Revision Anterior Cruciate Ligament Reconstruction
- Control Arm (Sham Comparator): Patients undergoing revision anterior cruciate ligament reconstruction surgery will get a sham incision in lieu of bone marrow harvesting.
  Interventions: Procedure: Sham Incision; Procedure: Revision Anterior Cruciate Ligament Reconstruction

INTERVENTIONS:
Biological: Concentrated Bone Marrow Aspirate Injection — Intraoperatively, bone marrow will be harvested from the iliac crest with a commercial kit, it will then be prepared via centrifugation and an injection of the resulting concentrated product (cBMA) will be administered in the operative knee. cBMA is an autologous biologic product.
  Other Names: cBMA; BMAC; Bone Marrow Aspirate Concentrate
  Arms: Investigational Arm
Procedure: Sham Incision — A 2 mm sham incision will be made in the anatomical site where bone marrow would be harvested.
  Arms: Control Arm
Procedure: Revision Anterior Cruciate Ligament Reconstruction — This is the standard-of-care surgical procedure.
  Other Names: Revision ACLR

SUMMARY:
The goal of this pilot randomized clinical trial is to look into the efficacy of concentrated bone marrow aspirate (cBMA) in improving post traumatic osteoarthritis (PTOA) symptoms in patients undergoing revision anterior cruciate ligament reconstruction surgery. The main questions it aims to answer are whether clinical outcomes, such as pain, are improved in patients who get cBMA with surgery, if there is a change in circulating markers of inflammation and what part of the cellular and molecular composition of cBMA may explain its effects.

DETAILED DESCRIPTION:
Anterior cruciate ligament reconstruction (ACLR) surgery is considered a relatively safe and effective procedure, however, up to 18% of grafts will fail and require revision surgery. Some studies have shown that these patients may be at increased risk of worse clinical outcomes, including fast progression toward post-traumatic osteoarthritis (PTOA). This is likely in part due to the inflammatory environment created within the joint. Concentrated bone marrow aspirate (cBMA) is a regenerative medicine therapy that contains soluble factors and connective tissue progenitor cells which may have immunomodulatory and pro-regenerative potential. The use of this therapy in conjunction with standard of care surgical treatment may help reduce the inflammatory microenvironment inside the joint, therefore modifying the conditions that might lead to developing long term complications such as PTOA.

The investigators hypothesize that cBMA treatment at the time of revision ACLR may improve clinical outcomes at 1 year after surgery and reduce the risk of developing PTOA-associated symptoms.

Participants will be randomized to either get a cBMA injection (investigational arm) at the time of surgery or a placebo incision (control arm). Biological specimens (blood, urine, synovial fluid), imaging data, functional tests and patient reported clinical outcomes will be measured at different time points during the study, for up to two years after the surgery. This will allow the investigators to evaluate the effect of cBMA in clinical outcomes. Biological specimens will be analyzed using molecular biology techniques to determine their composition, including the concentration of cells and other inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age 18 to 55
* Previous unilateral ACLR (Anterior Cruciate Ligament Reconstruction) within the last 5 years, and identified as having experienced failure of the primary ACLR
* Scheduled to have a revision ACLR surgery, with any graft type (including patellar tendon, hamstring, quad or allograft)
* Able to complete all study procedures and participate in a standardized physical therapy program

Exclusion Criteria:

* History of inflammatory arthritis or joint sepsis
* Prior or concurrent total or sub-total meniscectomy
* Prior or present avascular necrosis of the index knee
* Oral or intra-articular corticosteroid injection within 3 months
* Hyaluronic acid or PRP (Platelet-Rich Plasma) injection within 6 months
* Use of duloxetine, doxycycline, indomethacin, glucosamine and/or chondroitin (ongoing or within 2 months)
* Any clinical or laboratory abnormality greater than grade 3 CTCAE, which in the view of the investigator, will compromise the participant's safety.
* Planned arthroplasty in the index knee

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in patient reported knee pain | Baseline, 6 weeks, 6 months, 12 months and 24 months post-operative
  The primary outcome measured for this study will be postoperative knee pain. This will be achieved using the Knee Injury and Osteoarthritis Outcome Score (KOOS) standardized questionnaire, which will be electronically delivered to participants at baseline and at 6-weeks, 6-months, 12-months and 24-months postoperatively. This questionnaire measures 42 items in a Likert scale for 5 different dimensions: pain, other symptoms, activities of daily living, function in sports and recreation and knee-related quality of life. The questionnaire is scored as a percentage from 0 to 100, with 0 representing extreme knee problems and 100 indicating no knee related symptoms, and therefore better outcomes.

SECONDARY OUTCOMES:
Expression of local inflammatory biomarkers | Baseline and 6 weeks post-operative
  Synovial fluid collected before and 6 weeks after surgery will be analyzed using ELISA panels, looking for expression and concentration of markers of inflammation (e.g. IL-1β, TNFα) and matrix remodeling (COMP, CTXII)
Concentration of circulating inflammatory biomarkers | Baseline, 6 weeks and 12 months post-operative
  Biological samples (urine and blood) will be collected intraoperatively, and at 6-weeks and 12-months post-operatively. Samples will be processed and analyzed using ELISA panels, looking for the circulating concentration of markers of inflammation (e.g. IL-1β, TNFα) and matrix remodeling (COMP, CTXII).
Change from baseline in cartilage morphology | Baseline, 12 months post-operative
  Proton density weighted fast-spin-echo images will be acquired to assess cartilage morphology preoperatively and at 12 months post-operatively. Findings will be scored using the MRI Osteoarthritis Knee Score (MOAKS), which establishes criteria for assessing lesion grade (from 0 - best to 3 - worst) in fourteen distinct subregions.
Change from baseline in articular cartilage relative proteoglycan content and collagen fibril organization | Baseline, 12 months postoperative
  Combined T1ρ-T2 quantitative MRI image acquisition protocol will help determine the changes in relative proteoglycan content and collagen fibril organization within the knee articular cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Otero, Ph.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Emory Orthopaedics & Spine Center, Atlanta, Georgia
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No